CLINICAL TRIAL: NCT05319171
Title: Performance of Currently Available traNscaTHEter Aortic Valve Platforms in Inoperable Patients With Pure Aortic regurgitatiON of a Native Valve. The PANTHEON International Project.
Acronym: PANTHEON
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Luca Testa, MD, PhD, Contract Professor of CArdiology, IRCCS Policlinico S. Donato
Other Study IDs: 12345
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TAVR — TAVR

SUMMARY:
* To investigate the performance of currently available THVs in terms of safety and efficacy
* To evaluate potential predictors of THV embolization or migration (TVEM)
* To assess the impact of TVEM on prognosis

ELIGIBILITY:
Inclusion Criteria:

* severe aortic regurgitation
* prohibitive surgical risk

Exclusion Criteria:

* surgical candidates

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: inoperable patients with severe aortic regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Overall mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico S. Donato, Milan, Italy, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poletti E, De Backer O, Scotti A, Costa G, Bruno F, Fiorina C, Buzzatti N, Latini A, Rudolph TK, van den Dorpel MMP, Brinkmann C, Patel KP, Panoulas V, Schofer J, Giordano A, Barbanti M, Regazzoli D, Taramasso M, Saia F, Baumbach A, Maisano F, Van Mieghem NM, Sondergaard L, Latib A, Amat Santos IJ, Bedogni F, Testa L. Transcatheter Aortic Valve Replacement for Pure Native Aortic Valve Regurgitation: The PANTHEON International Project. JACC Cardiovasc Interv. 2023 Aug 28;16(16):1974-1985. doi: 10.1016/j.jcin.2023.07.026. PMID 37648345